CLINICAL TRIAL: NCT07369141
Title: PREcision meDICine in Treatment in CardioVascular Disease
Acronym: PREDICT-CVD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PREDICT-CVD; No 101112022 (Other Grant/Funding Number: Innovative Health Initiative Joint Undertaking (IHI JU)); No 10088702 (Other Grant/Funding Number: UK Research and Innovation (UKRI)); NL 009912 (Other: Overzicht van Medisch-wetenschappelijk Onderzoek in Nederland (OMON))
Record Dates: First submitted 2025-12-31; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure; Acute Decompensated Heart Failure
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Proof of concept trial
Who Masked: Outcomes Assessor
Masking Description: Clinical endpoint committee remains blinded to allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard treatment for HF
  Interventions: Other: Standard of Care (Investigator Choice)
- Intervention (Experimental): AI algorithm to assist the treating HF professional in treatment decision
  Interventions: Other: ASSIST-HF AI- algorithm

INTERVENTIONS:
Other: ASSIST-HF AI- algorithm — AI-derived biomarker-guided treatment algorithm to assist the treating HF professional in treatment decision
  Arms: Intervention
Other: Standard of Care (Investigator Choice) — Standard treatment of care for HF
  Arms: Standard of Care

SUMMARY:
The main goal of PREDICT-CVS is to demonstrate that a personalized, AI-derived biomarker-guided medication treatment algorithm that provides advice to the treating professional is superior to prevent clinical events and improve quality of life (QoL) when compared to patients receiving standard treatment of care.

Participants will be randomized into two groups

* Group 1 - Standard treatment Participant will receive the usual treatment for heart failure, based on current medical guidelines.
* Group 2 - AI-supported treatment The professional will receive a personalized treatment plan generated by the AI program. This plan is based on medical information and biomarkers. The professional can choose whether or not to follow the AI's advice, reasons for not following the AI-based advice will be collected.

Participants will visit the outpatient clinic at 1, 2, 3 and 9 months after being randomized.

DETAILED DESCRIPTION:
The PREDICT-CVD is a prospective, randomized controlled, open label, multinational trial, in which patients with HF will be randomized to either the control arm or the intervention arm. The control arm is the standard of care and the intervention arm is where an AI-derived biomarker-guided treatment algorithm will be applied, to assist the treating professional in treatment decision. Assessment of the primary endpoint will be at the 9 month onsite follow-up visit, further long-term outcomes will be collected via telephone visits every 6 months until the last subject has completed the 9 month onsite follow-up.

The main objective is to demonstrate that a personalized, AI-derived biomarker-guided medication treatment algorithm that provides advice to the treating HF professional is superior to prevent clinical events and improve quality of life (QoL) when compared to patients receiving standard treatment of care.

The primary outcome of the trial is a clinical benefit, defined as a hierarchical composite of death from any cause, number of heart failure events and or a greater difference in change from baseline in the Kansas City Cardiomyopathy Questionnaire Total Symptom Score at 9 months, as assessed using a win ratio.

The expected duration for patients will be between 9 and max 24 months from the moment of enrollment. From 9 months onwards patients will be contacted by phone every 6 months and information regarding (HF) events and concomitant medication will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written and dated informed consent for participation prior to trial admission,
2. Age ≥18 years, female or male
3. Diagnosis of heart failure* either before discharge of a heart failure hospital admission or in the outpatient setting,
4. Symptomatic, defined as NYHA class II - IV,
5. LVEF < 50% measured in the last 12 months (using any modality), with no occurrence of HF event(s) since that measurement) and
6. Those not previously treated with evidence-based therapies or sub-optimally treated with GDMT defined as; • Not treated with one of the foundational four** HF medication unless absolute contraindication or documented intolerance

   * Definition of heart failure according to the most recent Heart Failure Guidelines of the European Society of Cardiology

     * Foundational four heart failure medication: BBs, ARNi, MRAs and SGLT2i. NB. This does not include ACE and ARBs these are permitted.

Exclusion Criteria:

1. Inability to understand and sign informed consent,
2. Scheduled or on renal replacement therapy,
3. Clearly documented intolerance to BBs, ARNI, SGLT2i or MRAs
4. Diagnosis of acute myocarditis or (non)obstructive hypertrophic cardiomyopathy,
5. The presence of a mechanical assist device,
6. Scheduled for mechanical assist device or heart transplant,
7. Acute coronary syndrome (ACS) in the past 3 months or current angina pectoris ≥class III,
8. Requiring valvular surgery or revascularization in the upcoming 3 months or revascularization within the past 3 months,
9. Anticipated need for surgery or any cardiovascular intervention, except implantable cardioverter defibrillator and/or cardiac resynchronization therapy, within 4 weeks,
10. Other non-cardiac conditions with limited life expectancy (≤ duration of the trial/ 1 year),
11. Participation in another (intervention) clinical trial (registry studies not included) until the onsite EoS visit (V5) at 9 months has been completed.
12. Women who are pregnant, breastfeeding or may be considering pregnancy during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit | 9 months
  Hierarchical composite of death from any cause, number of heart failure events and or a greater difference in change from baseline in the Kansas City Cardiomyopathy Questionnaire Total Symptom Score, as assessed using a win ratio

SECONDARY OUTCOMES:
Time to death from any cause | 9 months (the number of days/months from randomization to the date of death)
  time to the first (re)hospitalization due to disease progression
Time to first (re)-hospitalization due to heart failure | 9 months (the number of days/months from randomization to the date of first (re)-hospitalization due to heart failure)
  Time to first (re)-hospitalization due to heart failure
Time to all-cause hospitalization | 9 months (the number of days/months from randomization to the date of all cause hospitalization).
  Time to all-cause hospitalization
Time to cardiovascular (CV) mortality | 9 months (the number of days/months from randomization to the date of CV death)
  Time to cardiovascular (CV) mortality
Change in QoL | 9 months
  Change in QoL according to the KCCQ-TSS (change from baseline in KCCQ-TSS score, measured in points, with higher scores indicating better health status.)
Change in NT-proBNP | 9 months
  Change in NT-proBNP (pg/mL)
Change in clinical congestion score | 9 months
  Change in clinical congestion score (CCS). The higher the score the worst congestion is
Change in eGFR | 9 months
  Change in eGFR (mL/min/1.73 m²)
GDMT at 9 month | 9 months
  Guideline directed Medical Therapy

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided
not decided at this time yet